CLINICAL TRIAL: NCT01030497
Title: Feasibility Study for Detection of Cervical Lymph Node Metastases With a High-Resolution PET Imaging System in Patients With Known or Suspected Cancers of the Upper Aerodigestive Tract
Brief Title: Detection of Cervical Lymph Node Metastases With a High-Resolution Positron Emission Tomography (PET) Imaging System
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0477
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Head and Neck Cancer
Keywords: Cancer; Cervical Lymph Node Metastases; High-Resolution PET Imaging System; Upper Aerodigestive Tract; Head; Neck; HR PET Imaging System; High-Resolution PET; PET/CT; PEMFlex Solo II; positron emission tomography/computed tomography (PET/CT)
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this clinical research study is to learn if using the PEMFlex Solo II, a high-resolution camera for PET scan imaging, on an area of the body that has, or is suspected to have cancer will give researchers the same or better information about the disease compared to the images taken with a routine PET/CT.

Researchers will compare the images taken using the PEMFlex Solo II to the images taken during your scheduled routine PET/CT scan, as well as any additional routine CT scan(s), magnetic resonance imaging (MRI) scan(s), and/or ultrasound image(s) you may have had within the last 30 days or may have in the next 30 days.

DETAILED DESCRIPTION:
If you agree to take part in this study, right after your already scheduled routine PET/CT scan is complete, a study staff member will take you to a separate imaging room located in the same clinic area where your routine PET/CT scan was just performed.

You will then sit in a chair as a study staff member positions the PEMFlex Solo II on either side of the part of the neck that has, or is suspected to have cancer. It will take about 20 minutes to set up the PEMFlex Solo II and take the PET scan images.

Length of Study:

After the PET scan images have been taken using the PEMFlex Solo II, your participation in this study will be over.

This is an investigational study. The PEMFlex Solo II is commercially available for PET scan imaging of the breast. Using the PEMFlex Solo II for imaging any other parts of the body is investigational.

Up to 10 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent.
2. Known or suspected primary cancer of the upper aerodigestive tract, which may be determined by biopsy, physical examination- including upper endoscopy or noninvasive imaging studies including CT, MR, ultrasound, or prior PET.
3. Known or suspected metastatic disease to cervical lymph nodes based on physical examination, imaging studies or biopsy.
4. Scheduled for routine clinical imaging at the ACB PET/CT facility.
5. Participant must be at least 18 years of age.

Exclusion Criteria:

1. Prior treatment (chemotherapy, radiotherapy) for cancer of the upper aerodigestive tract.
2. Prior biopsy procedures, including resection of the primary cancer, will not exclude the patient from participation.
3. Uncontrolled blood glucose levels (>200 mg/dl).
4. Patient is unable to comprehend the requirements of the study.
5. Patient is unable to undergo scanning of the neck with the PEM (PET) scanner (due to body habitus, inability to comply with positioning requirements, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected primary cancer of the upper aerodigestive tract or metastatic disease to cervical lymph nodes, over 18 years of age, and scheduled for routine clinical imaging at the PET/CT facility.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of peripheral tumor lesions identified in standard PET/CT imaging also identifiable in PEM images. | 20 minutes for imaging using PEMFlex Solo II, within ± 30 days of standard PET/CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rohren, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org